CLINICAL TRIAL: NCT01851278
Title: Effectiveness and Tolerance Infiltration Intraarticular Corticosteroid According to Dose
Brief Title: Effectiveness Intraarticular Corticosteroid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Daniele Freitas Pereira, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIA- 3131- AR
Record Dates: First submitted 2013-04-12; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: injection; arthritis; corticosteroid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose (Active Comparator): intraarticular wrist injection of 40mg, 2ml
  Interventions: Drug: Triamcinolone hexacetonide
- low dose (Active Comparator): intraarticular wrist injection of 20mg, 1ml.
  Interventions: Drug: Triamcinolone hexacetonide

INTERVENTIONS:
Drug: Triamcinolone hexacetonide — High dose means 40mg or 2ml of triamcinolone hexacetonide
  Arms: high dose
Drug: Triamcinolone hexacetonide — Low dose means 20mg or 1 ml of triamcinolone hexacetonide
  Arms: low dose

SUMMARY:
The purpose of this study is to compare the small and large dose of corticosteroid used in intraarticular injection of wrist.

DETAILED DESCRIPTION:
Background / Objectives: The optimal dose of corticosteroid to be used in intraarticular injection is not well established. The objective of this study is to compare the effectiveness and tolerance in the medium-term between small and large dose of triamcinolone hexacetonide (TH) used in intraarticular injection (IAI) of medium size joint of patients with rheumatoid arthritis (RA). Materials/Methods: A controlled, randomized, prospective, double-blind study will be realized in patients with RA. It will be evaluated 60 wrists joints (representing medium size joints) from the outpatient clinics at the Rheumatology Division UNIFESP, Brazil. Inclusion criteria were: patients with established RA, age between 18 and 65 years, disease modifying anti-rheumatic drugs (DMARDs) stable for at least 3 months, synovitis in wrist with pain visual analogic scale (VAS) between 4 and 8cm. Patients with overlap syndromes, polyarticular synovitis, diabetes mellitus or uncontrolled hypertension and those with suspected local or systemic infection were excluded. Patients will be randomized (Clapboard randomization) in two groups of 30 patients each: group 1 (high dose) is injected with 40mg (2ml) of TH and group 2 (small dose) was injected 20mg (1ml). Only one joint is injected by patient (IAI blindly). Evaluation will be conducted by a blinded observer at five times: baseline (T0), one week (T1), four (T4), eight (T8) and twelve (T12) weeks and the following assessment instruments were used: visual analogue scale for pain and swollen (VAS 0-10cm); wrist goniometry; chronic disease activity index (CDAI). Side effects and related events were reported in a medical questionnaire. The level of statistical significance was 5%.

ELIGIBILITY:
Inclusion Criteria:

* patients with established RA
* age between 18 and 65 years
* disease modifying anti-rheumatic drugs (DMARDs) stable for at least 3 months
* synovitis in wrist with pain visual analogic scale (VAS) between 4 and 8cm

Exclusion Criteria:

* patients with overlap syndromes
* polyarticular synovitis
* diabetes mellitus or uncontrolled hypertension and those with suspected local or systemic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-10 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | up to 12 weeks

SECONDARY OUTCOMES:
chronic disease activity index (CDAI) | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniele F Pereira, MsC, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Universidade Federal de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Konai MS, Vilar Furtado RN, Dos Santos MF, Natour J. Monoarticular corticosteroid injection versus systemic administration in the treatment of rheumatoid arthritis patients: a randomized double-blind controlled study. Clin Exp Rheumatol. 2009 Mar-Apr;27(2):214-21. PMID 19473560